CLINICAL TRIAL: NCT03334799
Title: A Case-Control Pilot Study on the Biomechanical Effects of Wearing a Sacroiliac Belt in Women
Brief Title: Biomechanical Effects of Wearing a Sacroiliac Belt in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 14-2323
Record Dates: First submitted 2017-10-24; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Pelvic Girdle Pain
Keywords: sacroiliac belt; kinematics; stability; pelvic girdle pain; sacroiliac instability
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Intervention Model Description: case control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacroiliac belt on and off (Other): Belt on and belt off
  Interventions: Device: sacroiliac belt

INTERVENTIONS:
Device: sacroiliac belt — standing and walking with the belt on and with the belt off
  Other Names: pelvic belt

SUMMARY:
Women with pelvic girdle pain PGP) often get relief from using a sacroiliac belt. The study will explore if there are differences and in the changes of lower body movement in stability with the belt on and with the belt off. Women with PGP will be matched with women without to explore if there is a difference between these two groups. This will be looked at in standing and in walking.

DETAILED DESCRIPTION:
SacroIliac (SI) joint dysfunction (also called pelvic girdle pain) has been associated with impaired load transfer across the lumbopelvic region. This can result in lower back pain as well as poor biomechanical adaptation during walking. Sacroiliac (SI) belts have typically been prescribed in order to mitigate pain and improve load transfer in individuals with SI joint dysfunction. It has been speculated that SI belts have the ability to instantaneously increase joint stability, and as a result improve load transfer and muscle activation and recruitment. However, this speculation is primarily based on anecdotal evidence; there is little biomechanical research supporting the effects of wearing an SI belt. In order to gain an improved understanding of the biomechanical effects of wearing an SI belt, the investigators propose to conduct a study with the following key objectives:

1. Determine if there are differences with respect to neuromuscular, kinematic, or pressure patterns during walking and/or standing between healthy stable individuals and individuals with SI joint dysfunction
2. Determine if wearing an SI belt affects neuromuscular, kinematic, or pressure patterns during walking and/or standing in women with sacroiliac instability

Variables measured will include:

1. Kinematics will be collected to quantify posture and joint angles
2. Kinetics will be collected to quantify ground reaction forces
3. Plantar pressure will be collected to quantify force distribution and center or pressure
4. Joint moments (Lumbar-pelvic and Hip) will be added as variables. The investigators will use inverse dynamics to calculate various joint moments during walking.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Individuals with isolated SI joint dysfunction
* Individuals with shoe size 6, 7, 8 or 9 US

and matched controls by age (within 5 years), BMI (within one point) and parity

Exclusion Criteria:

* Pregnancy in the last year or presently pregnant
* Significant lumbar dysfunction
* Significant hip dysfunction
* Leg length discrepancy of 1 cm or more
* Women who have previously undergone prolotherapy or SI joint injections
* Women with previous lower back, hip, knee or ankle surgery
* Inability to stand for 60 sec unaided or to walk unaided.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 10 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2017-09-09 (Actual)

PRIMARY OUTCOMES:
Explore if 95% confidence ellipse area of the center of pressure or kinematic measures can distinguish women with PGP from women without PGP when a SI belt is applied | within 2 months of enrollment, measured at one point in time
  Pressure insoles will be used to quantify the 95% confidence ellipse area of the CoP determined from each of the 2 feet, during the 30 second standing trials. The sampling will be compounded at a rate of 100 Hz and provided a time-pressure series with a range from 15 to 1200 kPa. The 95% confidence ellipse area of both feet will be summed. The average of the 3 trials will be used. Kinematic data will be collected using eight high speed video cameras at a sample rate of 240 Hz. All test subjects will be equipped with a marker set consisting of 32 light reflecting markers according to Visual3D (C-Motion, Inc., Germantown, USA) marker set guidelines. All measurements will be made on the right side. Walking speed will be monitored using photo electronic cells. Identified and averaged for 10 over-ground walking trials for each participant using custom Matlab software (MathWorks Inc., Natick, MA, USA).

SECONDARY OUTCOMES:
95% confidence ellipse area of the center of pressure | within 2 months of enrollment, measured at one point in time
  Pressure insoles (Pedar, novel GmbH, Germany) will be used to quantify the 95% confidence ellipse area of the CoP determined from each of the 2 feet, during the 30 second standing trials. The sampling will be compounded at a rate of 100 Hz and provided a time-pressure series with a range from 15 to 1200 kPa. Prior to testing, the insoles will be calibrated as per the manufacture's protocol. All data will be analyzed using custom Matlab scripts. The 95% confidence ellipse area of both feet will be summed. The average of the 3 trials will be used.Gait variability will be assessed by calculating the average position of the CoP in the medial-lateral direction during walking using pedar pressure insoles. The mean and standard deviation of the average CoP position will be defined as gait variability in medial-lateral direction calculated for each subject, foot, and condition.
kinematic changes of lower extremity | within 2 months of enrollment, measured at one point in time
  A force plate (Kistler Instrumente AG, Switzerland) recording at 2400 Hz will be positioned in the middle of a 15 meter walkway to measure ground reaction forces (GRF) during standing and walking. The threshold for determining heel strike wil be 20 N. Walking speed will be monitored using photo electronic cells (model TC Timing System; Brower Timing Systems, Draper, UT). Discrete kinematic and kinetic variables will be identified and averaged for 10 over-ground walking trials for each participant using custom Matlab software (MathWorks Inc., Natick, MA, USA).
  Kinematic data will be collected using eight high speed video cameras (Motion Analysis Corporation, Santa Rosa, USA) Version 3.6.1.1315 at a sample rate of 240 Hz. All test subjects will be equipped with a marker set consisting of 32 light reflecting markers according to Visual3D (C-Motion, Inc., Germantown, USA) marker set guidelines. All measurements will be made on the right side.

CONTACTS AND LOCATIONS:
Overall Officials: Magali Robert, Principal Investigator — Foothils Hospital Cumming School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided
Data will be stored in repository for access by request